CLINICAL TRIAL: NCT05572138
Title: Body Impedance Analysis to Detect Muscle Strength Associated With ICU Acquired Weakness
Brief Title: Body Impedance Analysis to Detect ICUAW
Acronym: BIAMI
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Stefan J Schaller, Deputy Clinical Director, Charite University, Berlin, Germany
Other Study IDs: BIAMI
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients
  Interventions: Diagnostic Test: Body Impedance Analysis

INTERVENTIONS:
Diagnostic Test: Body Impedance Analysis — Body Impedance Analysis

SUMMARY:
The aim of the study is to detect a value of muscle and organ mass measured by body impedance analysis and its correlation with the Medical Research Council (MRC) score. An MRC score ≤ 48 is defined as a diagnosis of ICU acquired weakness. The correlation of the values detected by BIA and their transfer to an MRC Score ≤ 48 will be investigated.

The knowledge gained will be used for early detection of ICUAW in order to reduce the consequences of the same.

DETAILED DESCRIPTION:
Intensive Care Unit Acquired Weakness (ICUAW) describes the clinically diagnosed manifestation of neuromuscular organ dysfunction. It develops in approximately 40% of all ICU patients, which corresponds to at least 1.2 million patients annually in Germany. All these patients face a wide spectrum of sequelae and increased mortality up to 5 years after ICU discharge. A characteristic pathophysiological phenomenon is early severe muscle atrophy, which is as high as 17% in the first days after ICU admission.

ICUAW is currently diagnosed by the MRC score, which is assessed by the sum of manual muscle strength test results in 12 muscle groups (sum score). Manual muscle testing (MMT) is not possible during the early phase in critical illness in most patients due to coma, delirium, and/or injury. In addition, there is a possible discrepancy by different observers. As a result, early detection of ICUAW may be inadequate in most patients and unreliable during critical illness.

Measurement by BIA is reproducible, so differences in measurement can be attributed to changes in clinical condition. Body impedance analysis thus demonstrates a means of objective measurement.

Thus, the study aims to counteract the long-term consequences of ICUAW through early detection of ICUAW by allowing countermeasures to be taken earlier.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged ≥ 18 years with ventilatory support within 36 hours from ICU admission.

Exclusion Criteria:

* With a language barrier
* Patients with pacemaker or other electronic implant
* Expected death or discontinuation of life-sustaining measures.
* Not walking independently before hospitalization (gait aids allowed)
* Allergy to electrode gel
* BIA or ultrasound not technically feasible due to e.g. extensive wounds, skin rash or bandages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill invasively ventilated patients
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-01-28 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
Correlation: Skeletal muscle mass and MRC-Score | till Day 30
  The primary endpoint is the correlation between Skeletal muscle mass (SMM) measured by BIA and MRC score.

SECONDARY OUTCOMES:
Correlation CSA and Skeletal muscle mass | till Day 30
  Cross sectional area of muscle ultrasound (M. rectus femoris) and Skeletal muscle mass (SMM) measured by BIA
UCR : MRC correlation | till Day 30
  Correlation of urea-creatinine ratio in blood with MRC score.
Kreatinin : MRC correlation | till Day 30
  Correlation of creatinine in blood with MRC score.
IMS during the ICU stay | till Day 30 or ICU discharge
  achieved mobilization level during the ICU stay using the ICU Mobility Scale (IMS)
ICU mortality | till Day 30
  Mortality during ICU stay
Duration of Mechanical ventilation | till Day 30
  Duration of invasive mechanical ventilator dependency
Hospital mortality | till Day 30
  Mortality during Hospital stay
ICU-LOS | till Day 30 (till ICU discharge)
  Length of stay in the ICU
Hospital LOS | till Day 30 (till hospital discharge)
  Length of stay in the hospital
in-hospital mortality | till Day 30 (till hospital discharge)
  Mortality during the Hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Stefan J Schaller, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Univiversitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Background] Kyle UG, Bosaeus I, De Lorenzo AD, Deurenberg P, Elia M, Gomez JM, Heitmann BL, Kent-Smith L, Melchior JC, Pirlich M, Scharfetter H, Schols AM, Pichard C; Composition of the ESPEN Working Group. Bioelectrical impedance analysis--part I: review of principles and methods. Clin Nutr. 2004 Oct;23(5):1226-43. doi: 10.1016/j.clnu.2004.06.004. PMID 15380917
- [Background] Savalle M, Gillaizeau F, Maruani G, Puymirat E, Bellenfant F, Houillier P, Fagon JY, Faisy C. Assessment of body cell mass at bedside in critically ill patients. Am J Physiol Endocrinol Metab. 2012 Aug 1;303(3):E389-96. doi: 10.1152/ajpendo.00502.2011. Epub 2012 May 29. PMID 22649067
- [Background] Fan E, Cheek F, Chlan L, Gosselink R, Hart N, Herridge MS, Hopkins RO, Hough CL, Kress JP, Latronico N, Moss M, Needham DM, Rich MM, Stevens RD, Wilson KC, Winkelman C, Zochodne DW, Ali NA; ATS Committee on ICU-acquired Weakness in Adults; American Thoracic Society. An official American Thoracic Society Clinical Practice guideline: the diagnosis of intensive care unit-acquired weakness in adults. Am J Respir Crit Care Med. 2014 Dec 15;190(12):1437-46. doi: 10.1164/rccm.201411-2011ST. PMID 25496103
- [Background] Appleton RT, Kinsella J, Quasim T. The incidence of intensive care unit-acquired weakness syndromes: A systematic review. J Intensive Care Soc. 2015 May;16(2):126-136. doi: 10.1177/1751143714563016. Epub 2014 Dec 18. PMID 28979394
- [Background] Van Aerde N, Meersseman P, Debaveye Y, Wilmer A, Gunst J, Casaer MP, Bruyninckx F, Wouters PJ, Gosselink R, Van den Berghe G, Hermans G. Five-year impact of ICU-acquired neuromuscular complications: a prospective, observational study. Intensive Care Med. 2020 Jun;46(6):1184-1193. doi: 10.1007/s00134-020-05927-5. Epub 2020 Jan 22. PMID 31970446
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Wollersheim T, Woehlecke J, Krebs M, Hamati J, Lodka D, Luther-Schroeder A, Langhans C, Haas K, Radtke T, Kleber C, Spies C, Labeit S, Schuelke M, Spuler S, Spranger J, Weber-Carstens S, Fielitz J. Dynamics of myosin degradation in intensive care unit-acquired weakness during severe critical illness. Intensive Care Med. 2014 Apr;40(4):528-38. doi: 10.1007/s00134-014-3224-9. Epub 2014 Feb 15. PMID 24531339
- [Background] Hough CL, Lieu BK, Caldwell ES. Manual muscle strength testing of critically ill patients: feasibility and interobserver agreement. Crit Care. 2011;15(1):R43. doi: 10.1186/cc10005. Epub 2011 Jan 28. PMID 21276225
- [Background] Gijsen M, Simons E, De Cock P, L N G Malbrain M, Wauters J, Spriet I. Reproducibility of fluid status measured by bioelectrical impedance analysis in healthy volunteers: a key requirement to monitor fluid status in the intensive care unit. Anaesthesiol Intensive Ther. 2021;53(3):193-199. doi: 10.5114/ait.2021.105826. PMID 34284553
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328